CLINICAL TRIAL: NCT00250549
Title: A Randomized Control Trial Evaluating the Educational Effectiveness of a Rapid HIV Post-Test Counseling Video.
Brief Title: A Theory Based HIV Prevention Video For Rapid HIV Testing: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Bronx Healthcare Network (Other)
Responsible Party: Principal Investigator, Yvette Calderon,MD, MS, Professor of Clinical Emergency Medicine, North Bronx Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-190
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: HIV
Keywords: HIV; Prevention; Rapid HIV testing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV counselor (No Intervention): Patients who tested for HIV and consent to participate in the study receive a posttest educational session with an HIV counselor. Afterwards, patients complete an assessment tool concerning HIV prevention and transmission.
- Post test video (Experimental): Patients who tested for HIV and consent to participate in the study watch a a 15-minute HIV posttest educational video available in English/Spanish. Afterwards, patients complete an assessment tool concerning HIV prevention and transmission.
  Interventions: Behavioral: Post test video

INTERVENTIONS:
Behavioral: Post test video — We compared the educational effectiveness of a 15-minute posttest counseling video with the normal practice of a session with an HIV counselor.Patients in the experimental group watched an HIV posttest educational video.
  Arms: Post test video

SUMMARY:
OraQuick is a safe, rapid test that accurately identifies HIV in as little as 20 minutes. By providing an accurate, quick method for detecting a person's serostatus and access to immediate post-test counseling, rapid testing has a crucial role in identifying HIV status and improving post-test counseling rates in populations who are at high risk of HIV infection and high failure to return rates. This prospective randomized control trial compared the educational effectiveness of a fifteen-minute post-test counseling video with the normal practice of a session with an HIV counselor.

DETAILED DESCRIPTION:
A convenience sample of stable patients presenting to the walk-in section of the Jacobi Medical Center Adult ED were recruited for rapid HIV testing. After consenting for the rapid HIV test and completing measures on condom intention and condom use self-efficacy, participants were randomized to either a fifteen-minute HIV post-test educational video available in English or to an HIV counselor for post-test counseling. Afterwards, both groups completed a measure of HIV knowledge assessing relevant testing information and level of satisfaction. An equivalence analysis was carried out to assess whether the video was at least as good as counseling, measured by total score on the knowledge questionnaire, with a lower equivalence bound of -5%.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients presenting to the Urgent Care Area at Jacobi Medical Center

Exclusion Criteria:

* Patients that were in to much pain, unable to understand the consent process or spoke another language other than the languages offered via the video or were HIV tested with in 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-05; Primary Completion 2005-10 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Mean Knowledge Score within both groups. | One year

SECONDARY OUTCOMES:
Overall condom intention measures and Condom Self efficacy measures | One year

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD, MS, Principal Investigator — Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States